CLINICAL TRIAL: NCT01649830
Title: Efficacy of Post-radiation Adjuvant Temozolomide Chemotherapy in Residue Low-grade Glioma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Zhongping Chen, Professor and Chair, Department of Neurosurgery, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012012
Record Dates: First submitted 2012-07-20; First posted 2012-07-25 (Estimated); Last update posted 2020-05-28 (Actual); Status verified 2020-05

CONDITIONS: Astrocytoma; Oligodendroglioma; Oligodendroastrocytoma
Keywords: low-grade glioma; radiotherapy; chemotherapy
MeSH Terms: conditions — Astrocytoma; Oligodendroglioma | interventions — Radiotherapy; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Radiotherapy plus adjuvant temozolomide (Experimental): Radiation therapy will start within 8 weeks after neurosurgical procedures. The residue gliomas will receive a total dose of 54.0 Gy in 27 - 30 fractions over 6 - 7 weeks. Four weeks after radiotherapy, patients will then receive 6 cycle of temozolomide dosed at 200 mg/m2 (150 mg/m2 for the first cycle) daily for 5 consecutive days, repeated every 28 days.
  Interventions: Radiation: Radiotherapy; Drug: Temozolomide
- Radiotherapy (Active Comparator): Radiation therapy will start within 8 weeks after neurosurgical procedures. The residue gliomas will receive a total dose of 54.0 Gy in 27 - 30 fractions over 6 - 7 weeks.
  Interventions: Radiation: Radiotherapy

INTERVENTIONS:
Radiation: Radiotherapy — External beam radiation: 54.0 Gy in 27 - 30 fractions over 6 - 7 weeks.
Drug: Temozolomide — dosed at 200 mg/m2 (150 mg/m2 for the first cycle) daily for 5 consecutive days, repeated every 28 days.
  Arms: Radiotherapy plus adjuvant temozolomide

SUMMARY:
Low-grade glioma (LGG) is a common primary brain tumor in young adults. The infiltrative nature and frequent growth in eloquent area in brain often makes total resection impossible. Until now, no agreement has been achieved on the treatment of LGG without total resection. Post-radiation adjuvant temozolomide (TMZ) is currently the standard of care for high-grade gliomas. Radiotherapy or TMZ is recommended for the treatment of residue low-grade gliomas. However, the efficacy of combined radiotherapy with adjuvant TMZ for residue LGG remains to be defined. In this randomized controlled trial, the investigators will test the hypothesis that radiotherapy with subsequent TMZ chemotherapy is superior to improve the progression-free survival of patients with residue LGG without significant impairment to quality of life compared to radiotherapy alone.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 years to 60 years
* Incompletely resected supratentorial WHO II astrocytoma, oligodendroglioma or oligodendroastrocytoma
* Karnofsky Performance Score ≥ 60
* Adequate bone marrow, liver and renal function
* Ability of subject to understand character and individual consequences of the clinical trial
* Written informed consent

Exclusion Criteria:

* Refusal to participate the study
* Known hypersensitivity or contraindication to temozolomide
* Previous irradiation, prior radiosurgery or prior chemotherapy
* Pregnant or lactating females
* Malignant tumor other than brain tumor
* Contraindicated for MRI examination
* Unable to comply with the follow-up studies of this trial

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 290 (Estimated)
Dates: Start 2012-07; Primary Completion 2025-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 5 years

SECONDARY OUTCOMES:
Quality of life | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Zhong-ping CHEN, MD, PhD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China